CLINICAL TRIAL: NCT07231757
Title: The Recor Paradise System™ Hypertension Coverage With Evidence Development Study
Brief Title: The RADIANCE CED Study
Status: Recruiting | Type: Observational
Sponsor: ReCor Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RADIANCE CED
Record Dates: First submitted 2025-09-15; First posted 2025-11-17 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Cardiovascular Diseases; Vascular Diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Vascular Diseases | interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Exposure Group (uRDN + SOC): A procedure or device code for the Paradise™ ultrasound renal denervation system (uRDN) and medication records indicating receipt of blood pressure-lowering medications.
  Interventions: Device: Ultrasound Renal Denervation (Paradise™ Ultrasound Renal Denervation (uRDN) System)
- Comparator Group (SOC): Medication records indicating receipt of blood pressure-lowering medications.

INTERVENTIONS:
Device: Ultrasound Renal Denervation (Paradise™ Ultrasound Renal Denervation (uRDN) System) — A catheter-based system that delivers ultrasound energy to the renal sympathetic nerves.
  Other Names: Paradise™ ultrasound renal denervation system
  Groups: Exposure Group (uRDN + SOC)

SUMMARY:
The RADIANCE CED study is a prospective observational study designed to evaluate the long-term effectiveness of ultrasound renal denervation in lowering blood pressure among patients with uncontrolled hypertension. Data will be collected from electronic health records (EHRs) of Medicare-eligible patients to support generalizability of outcomes to the broader Medicare population. Individual hospital enrollment is not required for this study and IRB exemption has been received by sponsor.

ELIGIBILITY:
Common Inclusion Criteria:

* Adults aged ≥65 years with uncontrolled hypertension
* Stable regimen of blood pressure-lowering medication

Common Exclusion Criteria:

* Hypertension due to secondary causes
* Prior renal denervation treatment
* Pregnancy
* End-stage renal disease, dialysis, or kidney transplant

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults aged ≥ 65 years with uncontrolled hypertension
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment for Changes in Blood Pressure | November 2025 - December 2029

SECONDARY OUTCOMES:
Occurrence of Adverse Cardiovascular and Cerebrovascular Event | November 2025 - December 2029
Changes in Anti-Hypertensive Medication | November 2025 - December 2029

CONTACTS AND LOCATIONS:
Overall Officials: Megan Coylewright, MD, Principal Investigator — Essentia Health; Amir Kaki, MD, Principal Investigator — Ascension St. John Hospital
Locations (1):
- Henry Ford St. John Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available.